CLINICAL TRIAL: NCT02047279
Title: Left Atrium Reduction Versus no Left Atrium Reduction for Patients With Enlarged Left Atria and Persistent or Long Standing Persistent Atrial Fibrillation Undergoing Mitral Valve Surgery
Brief Title: Ablation and Left Atrium Reduction During Mitral Valve Surgery for Atrial Fibrillation
Acronym: ALARM-vs-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Alexander Bogachev-Prokophiev, PhD, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-04-31491
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Mitral valve
MeSH Terms: conditions — Atrial Fibrillation | interventions — Maze Procedure; Radiofrequency Ablation; Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MVS + maze (Active Comparator): Procedure: Maze procedure, mitral valve surgery
  The scheme of lesion pattern: "box" lesion + line to mitral valve + line from "box" to left atrial appendage. The ablation procedure was performed by using a dry bipolar radiofrequency ablation clamp.
  The left atrial appendage was excluded in all cases. For mitral regurgitation or stenosis, the procedures will be a valve repair in the majority of cases. For valves that are not amenable to repair, a valve replacement will be performed.
  Interventions: Procedure: maze procedure; Procedure: mitral valve surgery
- MVS + maze + LA reduction (Experimental): Procedure: maze procedure, mitral valve surgery, left atrial reduction
  The scheme of lesion pattern: "box" lesion + line to mitral valve + line from "box" to left atrial appendage. The ablation procedure was performed by using a dry bipolar radiofrequency ablation clamp.
  The left atrial appendage was excluded in all cases. For mitral regurgitation or stenosis, the procedures will be a valve repair in the majority of cases. For valves that are not amenable to repair, a valve replacement will be performed.
  The enlarged left atria are plicated (suture technique) between the left and right pulmonary vein down to the inferior end of left atrial incision on the half-moon shape.
  Interventions: Procedure: maze procedure; Procedure: mitral valve surgery; Procedure: left atrial reduction

INTERVENTIONS:
Procedure: maze procedure — The scheme of lesion pattern: "box" lesion + line to mitral valve + line from "box" to left atrial appendage. The ablation procedure was performed by using a dry bipolar radiofrequency ablation clamp. The left atrial appendage was excluded in all cases.
  Other Names: surgical ablation; radiofrequency ablation
Procedure: mitral valve surgery — For mitral regurgitation or stenosis, the procedures will be a valve repair in the majority of cases. For valves that are not amenable to repair, a valve replacement will be performed.
  Other Names: mitral valve repair; mitral velve replacement
Procedure: left atrial reduction — The enlarged left atria are plicated (suture technique) between the left and right pulmonary vein down to the inferior end of left atrial incision on the half-moon shape.
  Other Names: left atrial volume reduction
  Arms: MVS + maze + LA reduction

SUMMARY:
The purpose of this study is to estimate left atrial volume reduction surgery concomitant with the maze procedure and mitral valve repair/replacement in patients with atrial fibrillation with an enlarged left atria.

DETAILED DESCRIPTION:
The Cox-Maze procedure has been a gold standard for the treatment of atrial fibrillation. Success of the modified maze procedure after valvular operation with an enlarged left atria and persistent and longstanding persistent atrial fibrillation remains suboptimal. The question addressed was: In adults undergoing a maze procedure for atrial fibrillation does left atrial size reduction compared to maze surgery alone improve maze surgery success?

ELIGIBILITY:
Inclusion Criteria:

* Able to sign Informed Consent and Release of Medical Information forms
* Age ≥ 18 years
* Clinical indications for mitral valve surgery for organic mitral valve disease Note: May include need for surgical management of functional tricuspid regurgitation or patent foramen ovale. Surgical intervention may be performed via sternotomy or minimally invasive procedure.
* a) Persistent atrial fibrillation (AF) within 6 months prior to randomization, defined as non self-terminating AF lasting greater than 7 days but no more than one year, or lasting less than 7 days but necessitating pharmacologic or electrical cardioversion.

Duration of AF must be documented by medical history and Presence of AF must be documented by a direct electrocardiographic assessment within 6 months prior to randomization.

b) Longstanding persistent AF is defined as continuous AF of greater than one year duration.

Duration of AF must be documented by medical history and Presence of AF must be documented by a direct electrocardiographic assessment upon arrival in the OR.

* left atrial diameter > 65mm
* Able to use heart rhythm monitor

Exclusion Criteria:

* AF is paroxysmal
* AF without indication for mitral valve surgery
* Concomitant coronary artery bypass grafting (CABG), aortic arch or aortic valve procedure
* Previous catheter ablation for AF
* Redo cardiac surgery
* Left ventricle ejection fraction (LV EF) < 35%
* Life expectancy of less than one year
* Mental impairment or other conditions that may not allow subject to understand the nature, significance, and scope of study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation | 12 months

SECONDARY OUTCOMES:
Rate of significant adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Bogachev-Prokophiev, PhD, Principal Investigator — Meshalkin Research Institute of Pathology of Circulation
Locations (1):
- Novosibirsk State Research Institute of Circulation Pathology, Novosibirsk, Russia